CLINICAL TRIAL: NCT02972580
Title: Characterization of Clinical Skeletal and Cardiac Impairment in Carriers of Duchenne Muscular Dystrophy (DMD) and Becker Muscular Dystrophy (BMD)
Brief Title: Characterization of Clinical Skeletal and Cardiac Impairment in Carriers of DMD and BMD
Status: Active, not recruiting | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Parent Project Muscular Dystrophy (Other)
Responsible Party: Principal Investigator, May Ling Mah, Principal Investigator, Nationwide Children's Hospital
Other Study IDs: IRB16-00319
Record Dates: First submitted 2016-07-25; First posted 2016-11-23 (Estimated); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The blood sample for genetic testing will be delivered to the Molecular Genetics lab at Nationwide Children's Hospital, where genomic DNA will be isolated from peripheral white blood cells. DNA will be banked frozen while a portion of the sample will be delivered to the Emory Molecular Genetics Laboratories for testing of the DMD gene.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Cohort A: DMD/BMD Female Carriers who have/had an affected child (n=150)
  Interventions: Genetic: Genetic characterization
- Cohort B: DMD/BMD Female non-carriers controls who have/had an affected child (n=50)
  Interventions: Genetic: Genetic characterization
- Cohort C: Healthy Age-Matched Controls (n=50)
  Interventions: Genetic: Genetic characterization
- Cohort D: DMD/BMD Female Carriers with no affected children (n=25)
  Interventions: Genetic: Genetic characterization

INTERVENTIONS:
Genetic: Genetic characterization — Confirmatory genetic testing for mutation in DMD gene (Carrier Status) for subjects in respective Cohorts

SUMMARY:
Longitudinal prospective observational study. This is a 24-month study with the possibility of extending the data time points. Initially baseline, then 12 and 24 months follow up studies will be completed.

DETAILED DESCRIPTION:
Four cohorts are enrolled in this study. The target population is the cohort of genetically confirmed DMD/BMD female carriers (Cohort A). This cohort will consist of 150 DMD/BMD mothers who are somatic carriers of a mutation in the DMD gene. The data collected for this cohort will be compared to three control groups; Control Group B is a cohort of 50 DMD/BMD mothers who are NOT somatic carriers, Control Group C is a cohort of 50 age-matched healthy controls and Control Group D is a cohort of 25 genetically confirmed carriers who do not have an affected child. The inclusion of a Control Group B allows for a comparison to a group of mothers that share the emotional and cognitive burden of caring for an affected male without having the physical or cognitive risks of being a female carrier. The Control Group C offers robust data from an age-matched healthy cohort for purposes of comparison. Control Group D allows for comparison to a group of women that have the same physical or cognitive risks as the Cohort A female carriers, but do not have the same burden of care giving.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Cohort A requires a genetically confirmed mutation in the DMD gene with an affected child
* Cohort B includes DMD/BMD mothers with NO somatic mutation in the DMD gene
* Cohort C age-matched healthy controls with a normal CK level
* Cohort D requires a genetically confirmed mutation in the DMD gene without an affected child
* Able to complete testing in English
* Able to consent

Exclusion Criteria:

* Subjects with a contraindication to cardiac or skeletal muscle MRI
* Subjects on heart failure medication at time of enrollment
* Subjects on steroid treatment
* Presence of an inherited neurologic disease or comorbidity that may affect their ability to complete this study
* Has a medical condition or extenuating circumstance that, in the opinion of the investigator, might compromise the subject's ability to comply with the protocol required testing or procedures or compromise the subject's wellbeing, safety, or clinical interpretability

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort A: DMD/BMD Female Carriers who have/had an affected child (n=150) Cohort B: DMD/BMD Female non-carriers controls who have/had an affected child (n=50) Cohort C: Healthy Age-Matched Controls (n=50) Cohort D: DMD/BMD Female Carriers who do not have/had an affected child (n=25)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-06; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Compromise of cardiac function based on Cardiac Magnetic Resonance Imaging | 2 years
  Cardiac function as compromised by evidence of scarring of cardiac muscles, particularly of the base of the left ventricle via cardiac MRI studies with gadolinium contrast.

SECONDARY OUTCOMES:
Cardiac Function Assessment Treadmill SVO2 | 2 years
  Stress on heart muscle measured by SVO2 (percentage of oxygen saturation in the blood of the pulmonary artery). SVO2 represents an average of all the venous oxygen saturation of major organs and tissues. This measure provides assessment of cardiopulmonary function and helps measure the degree of cardiac instability and can be an indicator of deterioration from normal.
Physical Therapy Assessments Maximum Voluntary Isometric Contraction Testing | 2 Years
  MVICT measures strength of skeletal muscles by assessing the force generated by by individual muscles. The results can be compared to norms and deterioration can be assessed over time.
Physical Therapy Assessments 6 Minute Walk Test | 2 years
  A timed test to assess distance walked in 6 minutes is very quantitative and can be assessed in comparison to normal controls. Deterioration over time can be clearly measured.
Physical Therapy Assessments ACTIVE-seated | 2 Years
  Exploratory outcome quantifying upper extremity reaching ability using a custom-designed game telling how far the arm reaches in comparison to overall functional ability of the individual ability.
Physical Therapy Assessments Time-to-Rise | 2 Years
  A timed-test to measure ability to rise from the floor is quantifiable and measuring over time tells if there is loss of function.
Laboratory biomarkers - Creatine Kinase | 2 Years
  CK levels are an indicator of muscle breakdown.
Laboratory biomarkers - C-Reactive Protein | 2 Years
  Pro-inflammatory marker indicating the degree of inflammation of muscle when there is muscle breakdown.
Laboratory biomarkers - Interleukin-6 | 2 Years
  Pro-inflammatory marker indicating the degree of inflammation of muscle when there is muscle breakdown.
Laboratory biomarkers - Cortisol levels | 2 Years
  Hair cortisol levels measure stress levels as a means of understanding coping with disease.
Cognitive Assessment | 2 Years
  Cognitive function measured by Wechsler Abbreviated Scale of Intelligence (WASI) provides a possible tool to measure disease awareness and establish if IQ level correlates with disease-related stress.
Caregiver Stress | 2 Years
  Online self-report survey to assess stress burden on caregiver.
Pulmonary function testing (PFTs) | 2 Years
  Stable or improved FVC

CONTACTS AND LOCATIONS:
Overall Officials: May Ling Mah, MD, Principal Investigator — PI
Locations (1):
- Nationwide Children's Hosptial, Columbus, Ohio, United States

REFERENCES:
- [Derived] Mah ML, Cripe L, Slawinski MK, Al-Zaidy SA, Camino E, Lehman KJ, Jackson JL, Iammarino M, Miller N, Mendell JR, Hor KN. Duchenne and Becker muscular dystrophy carriers: Evidence of cardiomyopathy by exercise and cardiac MRI testing. Int J Cardiol. 2020 Oct 1;316:257-265. doi: 10.1016/j.ijcard.2020.05.052. Epub 2020 May 27. PMID 32473283